CLINICAL TRIAL: NCT04553003
Title: Glucocorticosteroid Therapy on Drug-induced Liver Injury: a Prospective Non-randomized Concurrent Control Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Yang (Other)
Responsible Party: Sponsor-Investigator, Li Yang, professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYang
Record Dates: First submitted 2020-08-30; First posted 2020-09-17 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Drug-induced Liver Injury
Keywords: glucocorticosteroid
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glucocorticoid+hepatoprotectant group (Experimental): glucocorticoid 0.4mg/kg/d+hepatoprotectant for 7d
  Interventions: Drug: Glucocorticoids+hepatoprotectant
- hepatoprotectant group (Active Comparator): hepatoprotectant for 7d
  Interventions: Drug: hepatoprotectant

INTERVENTIONS:
Drug: Glucocorticoids+hepatoprotectant — Participants received glucocorticoids (0.4mg/kg/d po.) and hepatoprotectant for 7 days.
  Other Names: prednisone; methylprednisolone
  Arms: glucocorticoid+hepatoprotectant group
Drug: hepatoprotectant — Participants received hepatoprotectants (i.v.gtt.) for 7 days.
  Other Names: Ademetionine1,4-Butanedisulfonate; Polyene Phosphatidyl choline
  Arms: hepatoprotectant group

SUMMARY:
The purpose of this study is to assess the safety and efficacy of glucocorticosteroid for treatment of drug-induced liver injury.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of DILI
2. RUCAM score≥6 and with liver histology
3. Meet any of the following conditions:

   1. TBIL ≥ 10 fold ULN ;
   2. TBIL ≥ 5 fold ULN and serum AST or ALT ≥ 20 fold ULN

Exclusion Criteria:

1. An chronic onset (≥6 months)
2. Other liver diseases, such as autoimmune liver diseases, viral hepatitis, etc
3. with contraindications of glucocorticoid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
percentage of patients that AST or ALT decline 25% at day 4 | Change from Baseline ALT and AST at day4
  AST or ALT decline 25% at day 4

SECONDARY OUTCOMES:
percentage of patients that AST or ALT decline 50% at day 8 | Change from Baseline ALT and AST at day8
  AST or ALT decline 25% at day 8
the time needed when TBIL decline 50% | up to 2 weeks
  TBIL decline 50%; time
incidence of side effects | up to 2 years
  infection，uncontrolled hypertension or hyperglycemia
relapse rate in 12 months after drug withdrawal | 12 months after drug withdrawal
  relapse rate
mortality in 12 months after drug withdrawal | 12 months after drug withdrawal
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology & Hepatology,West China Hospital,Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No